CLINICAL TRIAL: NCT01007240
Title: Clinical Study of the Antibacterial Properties of the Nano Particles Which Incorporated With the Soft Liner Silicone - in Obturators
Brief Title: Antibacterial Properties of Silicon Incorporated With Quaternary Ammonium Polyethylenimine Nanoparticles
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Dr Anat Sharon, Hadassah medical organization - maxillofacial rehabilitation department
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: siliconnanoHMO-CTIL
Record Dates: First submitted 2009-11-02; First posted 2009-11-04 (Estimated); Last update posted 2009-11-04 (Estimated); Status verified 2009-11

CONDITIONS: Carcinoma of Head and Neck
Keywords: head and neck carcinoma; obturators; maxillectomy; soft liner; nano particles; antibacterial properties; patients post maxillectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- soft liner with nano particles (Experimental): the obturators of this patients will be relined with soft liner, with incorporated nano particles. after a week, the soft liner will be taken off, and will be checked for bacterial adhesion.
  Interventions: Device: polyethylenimine (PEI) nanoparticles.

INTERVENTIONS:
Device: polyethylenimine (PEI) nanoparticles.

SUMMARY:
The aim of this study is to evaluate the antibacterial activity of crosslinked quaternary ammonium polyethylenimine (PEI) nanoparticles incorporated at 1-2% w/w in a commercial soft liner material when compared to the commercial soft liner material.

The investigators' results in vitro showed a significant delay in bacterial growth.

Therefore, the investigators assume to have the same delay in vivo- on patients.

ELIGIBILITY:
Inclusion Criteria:

* patients post maxillectomy, who are using obturators

Exclusion Criteria:

* patients who are not using obturators

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-05 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
bacterial growth | a week

CONTACTS AND LOCATIONS:
Overall Officials: anat b sharon, DMD, MSc, Principal Investigator — lecturer, department of maxillofacial rehabilitation, hadassah medical organiztion